CLINICAL TRIAL: NCT01118442
Title: Determination of the Acute Effects of Aortic Stenosis on Coronary Artery Haemodynamics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 1424
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Stenosis; Coronary Flow; Wave Intensity Analysis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myocardial biopsy specimens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Narrowing of the main valve which controls blood leaving the heart leads to a marked increase in death. To overcome this narrowing the heart muscle thickens abnormally and contracts more vigorously. However, in doing so, blood flow patterns to the heart muscle change through mechanisms which are incompletely understood. New technology allows such heart valve blockages to be fixed using balloons and metal stents inserted through tubes placed in arteries in the leg. Using sensors placed in these tubes it is possible to make detailed measurements of coronary flow and pressure, and apply new mathematical techniques to allow a better understanding of the detrimental effects that aortic stenosis has on coronary flow, before and after valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Severe Aortic Stenosis undergoing TAVI
* Normal coronary arteries
* Normal left ventricular function
* No other valvular pathology

Exclusion Criteria:

* Unable to consent
* Left ventricular impairment
* Left ventricular regional wall motion abnormality
* Other valve abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transcutaneous aortic valve insertion who meet study criteria
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2009-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Justin E Davies, MRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Davies JE, Sen S, Broyd C, Hadjiloizou N, Baksi J, Francis DP, Foale RA, Parker KH, Hughes AD, Chukwuemeka A, Casula R, Malik IS, Mikhail GW, Mayet J. Arterial pulse wave dynamics after percutaneous aortic valve replacement: fall in coronary diastolic suction with increasing heart rate as a basis for angina symptoms in aortic stenosis. Circulation. 2011 Oct 4;124(14):1565-72. doi: 10.1161/CIRCULATIONAHA.110.011916. Epub 2011 Sep 12. PMID 21911781